CLINICAL TRIAL: NCT00054561
Title: Phase III Randomized Study of Adjuvant Biologic Therapy in Patients With Stages III/IV Head and Neck Squamous Cell Carcinoma
Brief Title: Isotretinoin, Interferon Alfa, and Vitamin E in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000271174; ECOG-1301
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Interferon-alpha; Vitamin E; Isotretinoin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Dietary Supplement: vitamin E
Drug: isotretinoin
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as isotretinoin use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of tumor cells. Vitamin E may be able to decrease side effects caused by isotretinoin. It is not yet known whether combining isotretinoin and interferon alfa with vitamin E is more effective than observation in preventing recurrence of head and neck cancer after surgery and/or radiation therapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of isotretinoin and interferon alfa combined with vitamin E with that of observation in treating patients who have undergone surgery and/or radiation therapy for stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of adjuvant isotretinoin, interferon alfa, and vitamin E, in terms of incidence of primary disease recurrence and secondary primary tumor development, in patients with stage III or IV squamous cell carcinoma of the head and neck previously treated with definitive surgical excision and/or postoperative radiotherapy.
* Determine the qualitative and quantitative toxicity of this regimen in these patients.
* Compare the overall and disease-free survival of patients treated with this regimen vs those who undergo observation only.
* Determine whether alterations of p53 gene, retinoic acid receptors, retinoid-regulated gene, and interferon-responsive genes are associated with clinical outcome in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to T stage (T1 or T2 vs T3 or T4), N stage (N0 or N1 vs N2 or N3), prior therapy (complete tumor resection vs resection and radiotherapy/chemoradiotherapy vs radiotherapy or chemoradiotherapy alone), and prior chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral isotretinoin once daily, interferon alfa subcutaneously 3 times weekly, and oral vitamin E 3 times daily. Treatment repeats every month for 12 courses (1 year) in the absence of disease recurrence or unacceptable toxicity.
* Arm II: Patients undergo observation only for 1 year. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 376 patients (188 per treatment arm) will be accrued for this study within 3.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Primary site must be within the oral cavity, oropharynx, larynx, or hypopharynx
  * Stage III or IV primary lesion at diagnosis
  * No distant metastatic disease at diagnosis
  * No multiple primary lesions
* Currently disease-free after treatment with 1 of the following:

  * Complete tumor resection
  * Radiotherapy or chemoradiotherapy alone*
  * Resection followed by radiotherapy/chemoradiotherapy*
* No more than 4-16 weeks since prior surgery and/or radiotherapy/chemoradiotherapy NOTE: *Radiotherapy must have been 70-72 Gy in 1.8-2.0 Gy fractions to the primary tumor and clinically positive neck nodes and 44-50 Gy in 1.8-2.0 Gy fractions to clinically negative nodes, including the lower neck

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN

Renal

* Creatinine no greater than 1.2 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month prior to, during, and for 1 month after study therapy
* Electrolytes normal
* Fasting serum triglyceride level no greater than 2 times ULN (anti-triglyceride medication allowed)
* No other malignancy within the past 2 years except localized basal cell or squamous cell skin cancer
* No other concurrent medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered

  * Prior neoadjuvant chemotherapy allowed
  * Prior chemotherapy administered concurrently with radiotherapy allowed
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No history of megadose vitamin A (more than 25,000 I.U.)
* No other clinical trial enrollment that would preclude adjuvant systemic therapy
* No concurrent vitamin supplements containing vitamin A

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11-26 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong M. Shin, MD, Study Chair — Emory University
Locations (89):
- United States (82):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Burgess Health Center, Onawa, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Australia (2):
  - Westmead Breast Centre at NSW Breast Cancer Institute, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (3):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
  - San Juan City Hospital, San Juan
- Pretoria Academic Hospital, Pretoria, South Africa